CLINICAL TRIAL: NCT00766298
Title: Skeletal Muscle Lipid and Insulin Resistance: Effects of Physical Activity and Weight Loss
Acronym: SHELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Bret Goodpaster, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0406003
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Exercise; Weight Loss; Physical Activity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Weight Loss | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Weight Loss
  Interventions: Behavioral: Weight Loss
- 2 (Experimental): Exercise
  Interventions: Behavioral: Exercise
- 3 (Experimental): Exercise and Weight Loss
  Interventions: Behavioral: Exercise and weight loss

INTERVENTIONS:
Behavioral: Exercise — 16 week intervention; 6 exercise sessions weekly w 3 supervised exercise sessions weekly utilizing cycling or walking/jogging. Participants maintain exercise diaries: wks 1-4; 30 minutes at 60-70% MHR, wks 5-8; 40 minutes at 60-70% MHR, weeks 9-16; 40 minutes at 75% MHR
  Arms: 2
Behavioral: Weight Loss — The reduction of kcal/day through implementation of low fat diet
  Arms: 1
Behavioral: Exercise and weight loss — Exercise: 16 week intervention; 6 exercise sessions weekly w 3 supervised exercise sessions weekly utilizing cycling or walking/jogging. Participants maintain exercise diaries: wks 1-4; 30 minutes at 60-70% MHR, wks 5-8; 40 minutes at 60-70% MHR, weeks 9-16; 40 minutes at 75% MHR.
  Weight Loss: Reduction of kcal/day through implementation of a low fat diet.
  Arms: 3

SUMMARY:
102 late- life adults at risk for developing type 2 diabetes mellitus, will be randomized to one of three interventions designed to improve insulin sensitivity thereby potentially preventing future progression of type 2 diabetes. The investigators predict that insulin sensitivity will improve equally following either weight loss or exercise, while there will be additive effects from combined intervention.

The investigators hypothesize that weight loss will decrease intermuscular adipose tissue, intramyocellular lipid, and visceral abdominal adipose tissue.

DETAILED DESCRIPTION:
The primary objective of this project will be to examine the role of skeletal muscle lipid and capacity for fat oxidation in insulin resistance in older adults who either are at high risk for the development of type 2 diabetes mellitus (T2DM) or who are untreated newly diagnosed T2DM. A randomized intervention trial will be conducted to examine the effects of physical activity and weight loss, alone or in combination, on intramyocellular lipid (IMCL), intermuscular adipose tissue (IMAT) and abdominal AT (adipose tissue), oxidative capacity and insulin resistance.

The first aim is to examine the effects of weight loss without exercise on AT distribution, intramyocellular lipid (IMCL) and oxidative capacity of skeletal muscle in conjunction with improvements in insulin sensitivity. We will test the hypotheses that weight loss without exercise will: 1) Improve insulin sensitivity, decrease the lipid interspersed within muscle (intermuscular AT), intramyocellular lipid (IMCL), as well as visceral abdominal AT (VAT); and 2) Will have no effects on either skeletal muscle oxidative capacity determined in vitro or in vivo.

A second aim is to examine the effects of exercise without weight loss on AT, IMCL, oxidative capacity and insulin resistance. We will test the hypotheses that exercise without weight loss will: 1) Increase the oxidative enzyme capacity of muscle; 2) Increase IMCL despite having little effect on AT distribution within muscle (intermuscular AT) or visceral AT; 3) Improve insulin sensitivity to a similar degree as weight loss without exercise.

A third aim will be to examine the combined effects of exercise and weight loss on insulin resistance. Our third hypotheses are that combining weight loss and exercise will 1) Decrease IMAT, VAT and have little overall effect on IMCL 2) Improve the oxidative capacity of skeletal muscle; 3) Confer synergistic improvements in insulin sensitivity through the combined actions on AT and skeletal muscle capacity for oxidation.

A fourth aim will be to examine the combined effects of exercise and weight loss on subjects with newly diagnosed but untreated T2DM. Our final hypotheses are that exercise and weight loss will have similar effects in subjects with newly diagnosed T2DM compared to those at risk for developing T2DM with regards to improved insulin sensitivity, body composition and oxidative capacity of skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* 60-75 years of age
* Stable weight (No Gain/Loss of > 10 lbs in 6 months)
* Impaired Glucose Tolerance or Newly, untreated, undiagnosed type 2 diabetes
* Sedentary
* Non-smoker
* BMI 25.0-38.0 KG/M2
* Resting Blood Pressure ≤ 150mmHg systolic and ≤ 95 mmHg diastolic
* IGT: Fasting Glucose > 100, < 126 2-Hour OGTT > 140 but < 200
* T2D: Fasting Glucose > 126 < 2000 2-Hour OGTT > 200
* Note from PCP/Cardiologist for exercise clearance if positive stress test symptoms were observed from GXT

Exclusion Criteria:

* Clinically significant CVD including h/o MI
* Peripheral Vascular Disease
* Hepatic, renal, muscular/neuromuscular, or active hematologic/oncologic disease
* Clinically diminished pulse
* Presence of bruits in lower extremities
* Previous history of pulmonary emboli
* Peripheral Neuropathy
* Currently not engaged in a regular program and have a VO2 max pre-training value > 55 ml/kg-fat free mass-min., indicative of moderate fitness.
* Anemia (Hematocrit < 34%)
* Any contraindications to moderate exercise (Please specify)
* Inability and/ or unwillingness to comply with the protocol as written
* Active alcohol or substance abuse (Past 5 Years)
* Total cholesterol > 300 mg/dL
* Triglyceride > 350 mg/dL
* ALT > 80, AST > 80, Alk Phos > 240
* Proteinuria (defined as >1 + on routine dipstick), hypothyroidism (sTSH>8)
* Therapeutic Doses of Nicotinic Acid
* Oral glucocorticoids
* Females currently on hormone replacement therapy (HRT) less than 6 months
* Claustrophobia
* Previous difficulty with lidocaine or other local anesthetic
* Stress test symptoms:

  * Positive ECG (> 2mm ST segment depression) without PCP cardiologist permission to participate
  * Signs or symptoms of cardiovascular decomposition (hypotensive response to exercise)
  * Onset of angina or angina like symptoms, shortness of breath, change in heart rhythm, signs of poor perfusion (light-headedness), tightness,
  * Hypotension

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2004-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Effects of physical activity and weight loss, alone or in combination, on intramyocellular lipid, intermuscular adipose tissue and abdominal AT, oxidative capacity and insulin resistance. | 16 weeks

SECONDARY OUTCOMES:
Assess the mechanisms by which these interventions may prevent the development of diabetes | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bret H Goodpaster, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amati F, Dube JJ, Coen PM, Stefanovic-Racic M, Toledo FG, Goodpaster BH. Physical inactivity and obesity underlie the insulin resistance of aging. Diabetes Care. 2009 Aug;32(8):1547-9. doi: 10.2337/dc09-0267. Epub 2009 Apr 28. PMID 19401446
- [Result] Amati F, Dube JJ, Shay C, Goodpaster BH. Separate and combined effects of exercise training and weight loss on exercise efficiency and substrate oxidation. J Appl Physiol (1985). 2008 Sep;105(3):825-31. doi: 10.1152/japplphysiol.90384.2008. Epub 2008 Jul 10. PMID 18617627
- [Result] Amati F, Dube JJ, Stefanovic-Racic M, Toledo FG, Goodpaster BH. Improvements in insulin sensitivity are blunted by subclinical hypothyroidism. Med Sci Sports Exerc. 2009 Feb;41(2):265-9. doi: 10.1249/MSS.0b013e318187c010. PMID 19127201
- [Result] Amati F, Pennant M, Azuma K, Dube JJ, Toledo FG, Rossi AP, Kelley DE, Goodpaster BH. Lower thigh subcutaneous and higher visceral abdominal adipose tissue content both contribute to insulin resistance. Obesity (Silver Spring). 2012 May;20(5):1115-7. doi: 10.1038/oby.2011.401. Epub 2012 Jan 19. PMID 22262160
- [Result] Menshikova EV, Ritov VB, Fairfull L, Ferrell RE, Kelley DE, Goodpaster BH. Effects of exercise on mitochondrial content and function in aging human skeletal muscle. J Gerontol A Biol Sci Med Sci. 2006 Jun;61(6):534-40. doi: 10.1093/gerona/61.6.534. PMID 16799133
- [Derived] Dube JJ, Amati F, Toledo FG, Stefanovic-Racic M, Rossi A, Coen P, Goodpaster BH. Effects of weight loss and exercise on insulin resistance, and intramyocellular triacylglycerol, diacylglycerol and ceramide. Diabetologia. 2011 May;54(5):1147-56. doi: 10.1007/s00125-011-2065-0. Epub 2011 Feb 17. PMID 21327867